CLINICAL TRIAL: NCT05340205
Title: The Efficacy and Safety of Intrauterine Misoprostol Versus Intravenous Tranexamic Acid in Reducing Blood Loss During and After Cesarean Delivery in Patients With Placenta Previa: A Randomized Controlled Trial
Brief Title: Blood Loss During Cesarean Delivery in Placenta Previa Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noran Amin, Director, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Placenta previa disorders
Record Dates: First submitted 2022-04-11; First posted 2022-04-22 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa | interventions — Tranexamic Acid; Misoprostol; Oxytocin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tranexamic acid group (Active Comparator): Patients will receive 1 gm (10 ml) tranexamic acid diluted in 20 ml of Glucose 5% (administered as IV infusion over 5 minutes, at least 15 minutes prior to skin incision). Following the delivery of the baby, patients will additionally receive a slow IV bolus of 5 IU oxytocin and 20 IU oxytocin in 500 mL lactated Ringer's solution (infused at a rate of 125 mL/h).
  Interventions: Drug: Tranexamic acid
- Misoprostol group (Active Comparator): Patients will receive 400 microgram misoprostol which will be inserted inside the uterus near the cornu after delivery of the placenta and swabbing the uterine cavity. Patients will additionally receive a slow IV bolus of 5 IU oxytocin and 20 IU oxytocin in 500 mL lactated Ringer's solution (infused at a rate of 125 mL/h).
  Interventions: Drug: Misoprostol
- Oxytocin only (control) group (Active Comparator): Patients will receive only an IV bolus of 5 IU oxytocin and 20 IU oxytocin in 500 mL lactated Ringer's solution (infused at a rate of 125 mL/h) following the delivery of the baby.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Tranexamic acid — Patients will receive 1 gm tranexamic acid diluted in 20 ml of Glucose 5% 15 minutes prior to skin incision and a slow IV bolus of 5 IU oxytocin and 20 IU oxytocin in 500 mL lactated Ringer's solution (infused at a rate of 125 mL/h) following delivery of the baby.
  Other Names: Kapron
  Arms: Tranexamic acid group
Drug: Misoprostol — Patients will receive 400 microgram misoprostol which will be inserted inside the uterus near the cornu after delivery of the placenta and a slow IV bolus of 5 IU oxytocin and 20 IU oxytocin in 500 mL lactated Ringer's solution (infused at a rate of 125 mL/h).
  .
  Other Names: Cytotec
  Arms: Misoprostol group
Drug: Oxytocin — Patients will receive an IV bolus of 5 IU oxytocin and 20 IU oxytocin in 500 mL lactated Ringer's solution (infused at a rate of 125 mL/h) following the delivery of the baby.
  Other Names: Syntocinon
  Arms: Oxytocin only (control) group

SUMMARY:
To compare the efficacy and safety profile of intravenous tranexamic acid versus intrauterine misoprostol in reducing the blood loss during and after cesarean delivery in pregnant women diagnosed with placenta previa

DETAILED DESCRIPTION:
Placenta previa is defined as complete or partial covering of the internal os of the cervix with the placenta, at more than 16 weeks of gestation. It affects 0.3% to 2% of pregnancies in the third trimester and has become more evident secondary to the increasing rates of cesarean delivery (CD).

Placenta previa is a major risk factor for postpartum hemorrhage (PPH) and can lead to maternal and neonatal morbidity and mortality. Uncontrolled PPH from placenta previa may necessitate blood transfusion, hysterectomy, admission to the intensive care unit, or even death.

The efficacy of routine administration of oxytocin, to reduce the frequency of PPH after vaginal and cesarean birth is well-established. The Royal College of Obstetricians and Gynecologists recommends a slow IV bolus dose of 5 IU of oxytocin after delivery of the neonate in CD to ensure adequate uterine contractility, reduce intraoperative blood loss and prevent PPH. Likewise, the American College of Obstetricians and Gynecologists recommends the practice to use oxytocin but infusion instead of a bolus dose. Regardless of the mode of administration, oxytocin use in the setting of CD may result in maternal adverse effects, such as hypotension and tachycardia.

Misoprostol, a prostaglandin E1 analogue with strong uterotonic properties binds to myometrial cells to cause strong myometrial contractions. Misoprostol has been suggested as an alternative to injectable uterotonic agents for preventing PPH following vaginal or CD. It can be used orally, sublingually, buccally, rectally or put intrauterine with similar efficacy as oxytocin in reducing blood loss, preventing and treating PPH. Because of its availability, low cost, thermal stability, and ease of administration, misoprostol is suitable for worldwide use even in low resource settings in developing countries.

Tranexamic Acid (TA) is an analogue of lysine that inhibits fibrinolysis by competitively binding to plasminogen. It prevents the lysis of formed clot by inhibiting activation of plasminogen and plasmin. It is ten times more potent than amino-caproic acid. Several studies had assessed the use of TA in both the prophylaxis against and the treatment of PPH with the conclusion that TA reduces the following; blood loss in women with PPH, the need for hysterectomy, the risk of severe anemia and the need for further blood transfusion; hence, this could contribute significantly to the goal of reducing maternal mortality

ELIGIBILITY:
Inclusion Criteria:

* Parity: primigravida or multigravida.
* Gestational age: ≥ 36 weeks (confirmed by the first day of the last menstrual period or first trimester ultrasound scan).
* Candidate for termination of pregnancy by cesarean delivery.
* Singleton living healthy normally growing fetus.
* Cesarean delivery under spinal anesthesia.
* Pregnancies complicated with placenta previa diagnosed preoperatively by ultrasonography (placenta previa was defined as placenta partially or totally covers the cervix)

Exclusion Criteria:

* Patients diagnosed with morbidly adherent placenta.
* Placenta previa cases requiring cesarean hysterectomy in the primary surgery.
* Patients with preoperative anemia (Hemoglobin <9 gm/dl).
* History of thromboembolic event.
* Known allergy to tranexamic acid or prostaglandins.
* Bronchial asthma or other contraindications of misoprostol.
* Patients with other risk factors of postpartum hemorrhage (e.g., polyhydramnios, fetal macrosomia, uterine fibroid).
* Patients known to have bleeding tendency (e.g., those receiving anticoagulation, patients with thrombocytopenia, factor VIII or IX deficiency or Von Willebrand's disease).
* More than 2 previous cesarean deliveries procedures.
* Prolonged procedure (more than 2 hours from skin incision to skin closure).
* Concomitant maternal medical disorders (either chronic or pregnancy induced)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
To compare the estimated blood loss during cesarean delivery among the three groups | less than 2 hours
  The blood loss will be estimated in each of the three groups

SECONDARY OUTCOMES:
The Use of additional ecbolics denoting uterine atony | Baseline
  The need for extra ecbolics will be recorded
The occurrence of excessive blood loss (> 1000 mL) within the first 24 hours postoperatively | First 24 hours postoperatively
  Excessive blood loss will be recorded
The need for blood transfusion | During cesarean delivery and the first 24 hours postoperatively
  The need for blood transfusion will be recorded
The occurrence of any maternal side effects in the studied groups | First 6 hours postoperatively
  Maternal side effects will be recorded
The occurrence of any neonatal outcome in the studied groups | The first 6 hours postoperatively
  Neonatal side effects will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Tarek El Husseiny, MD, Study Director — Cairo University
Locations (1):
- Kasralainy Cairo University, Giza, Egypt

REFERENCES:
- [Background] Bhattacharya S, Ghosh S, Ray D, Mallik S, Laha A. Oxytocin administration during cesarean delivery: Randomized controlled trial to compare intravenous bolus with intravenous infusion regimen. J Anaesthesiol Clin Pharmacol. 2013 Jan;29(1):32-5. doi: 10.4103/0970-9185.105790. PMID 23493050
- [Background] Martinelli KG, Garcia EM, Santos Neto ETD, Gama SGND. Advanced maternal age and its association with placenta praevia and placental abruption: a meta-analysis. Cad Saude Publica. 2018 Feb 19;34(2):e00206116. doi: 10.1590/0102-311X00206116. PMID 29489954
- [Background] Prata N, Weidert K. Efficacy of misoprostol for the treatment of postpartum hemorrhage: current knowledge and implications for health care planning. Int J Womens Health. 2016 Jul 29;8:341-9. doi: 10.2147/IJWH.S89315. eCollection 2016. PMID 27536161
- [Background] Pabinger I, Fries D, Schochl H, Streif W, Toller W. Tranexamic acid for treatment and prophylaxis of bleeding and hyperfibrinolysis. Wien Klin Wochenschr. 2017 May;129(9-10):303-316. doi: 10.1007/s00508-017-1194-y. Epub 2017 Apr 21. PMID 28432428
- [Background] Sood AK, Singh S. Sublingual misoprostol to reduce blood loss at cesarean delivery. J Obstet Gynaecol India. 2012 Apr;62(2):162-7. doi: 10.1007/s13224-012-0168-2. Epub 2012 Jun 1. PMID 23543254
- [Background] Vogel JP, West HM, Dowswell T. Titrated oral misoprostol for augmenting labour to improve maternal and neonatal outcomes. Cochrane Database Syst Rev. 2013 Sep 23;2013(9):CD010648. doi: 10.1002/14651858.CD010648.pub2. PMID 24058051
- [Background] Della Corte L, Saccone G, Locci M, Carbone L, Raffone A, Giampaolino P, Ciardulli A, Berghella V, Zullo F. Tranexamic acid for treatment of primary postpartum hemorrhage after vaginal delivery: a systematic review and meta-analysis of randomized controlled trials. J Matern Fetal Neonatal Med. 2020 Mar;33(5):869-874. doi: 10.1080/14767058.2018.1500544. Epub 2018 Sep 10. PMID 30122082